CLINICAL TRIAL: NCT04371172
Title: The Impact of Transcatheter Aortic Valve Implantation on Cognition, Mood and Health-related Quality of Life - an Explorative Study
Brief Title: Impact of TAVI on Cognition, Mood and Health-related Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Andreas Baranyi, Prof., Medical University of Graz
Other Study IDs: 32-249 ex 19/20; 32-249 ex19/20 (Other: Ethikkommission, Medical university of Graz)
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with TAVI: cognitive research battery, MRI, laboratory values
  Interventions: Other: cognitive research battery, MRI, laboratory values

INTERVENTIONS:
Other: cognitive research battery, MRI, laboratory values — cognitive research battery, MRI, laboratory values

SUMMARY:
In the proposed study, patients with and without embolic protection devices during Transcatheter Aortic Valve Implantation will be repeatedly examined with a comprehensive psychiatric and cognitive test battery over a post-interventional period of 6 months after TAVI, with regard to the effects on mood, cognitive Performance and health-related Quality of life.

DETAILED DESCRIPTION:
The percutaneous aortic valve replacement (TAVI, Transcatheter Aortic Valve Implantation) enables the implantation of a new biological aortic valve at the beating heart. The procedure is performed under local anaesthesia and is a gold standard in the therapy of aortic stenosis, especially in patients with a too high health risk for cardiovascular surgery.

In the proposed study, patients with and without embolic protection devices during TAVI will be repeatedly examined with a comprehensive psychiatric and cognitive test battery over a post-interventional period of 6 months after TAVI, with regard to the effects on mood, cognitive Performance and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Written declaration of consent of the study participants to participate in the study after detailed information on the nature, significance, risks and scope of the study.
* Women and men between the ages of 19 and 90
* Clinical indication for TAVI intervention
* No previous psychiatric illness before TAVI
* No other serious disease affecting the immune system

Exclusion Criteria:

* Non-compliance with the inclusion criteria
* Persons unable to give consent (e.g. dementia, delirium etc.)
* Magnetic resonance imaging (MR) contraindications
* ophthalmological inability to read

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with percutaneous aortic valve replacement
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2025-05-29 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
cognition | 12 months
  Montreal-Cognitive-Assessment, cognitive test battery

SECONDARY OUTCOMES:
health-related quality of life | 12 months
  Short Form (36) Health Survey (SF-36): The SF-36 consists of 8 scales. scores. Each scale is directly transformed into a 0-100 scale. A score of 100 is equivalent to no disability.

OTHER OUTCOMES:
mood | 12 months
  Hospital Anxiety and Depression Scale (HADS): A person can score between 0 and 21 for either anxiety or depression); Montgomery-Åsberg Depression Rating Scale: usual cutoff points are: 0 to 6 - normal, 7 to 19 - mild depression, 20 to 34 - moderate depression, >34 - severe Depression
MRI | 12 months
  MRI

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baranyi, Prof., Principal Investigator — Medical University Graz, Austria
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided